CLINICAL TRIAL: NCT04030585
Title: Efficacy of Robot-assisted Exercise Program in Patients With Upper Limb Amputation Using Myoelectric Prosthesis
Brief Title: Robot-assisted Exercise in Patients With Amputation Using Myoelectric Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MYO-2019
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Prosthesis User; Amputation
Keywords: Amputation; robotic rehabilitation; Prosthesis
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Treatment group: robot-assisted exercise program Control: Home exercise program
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot-assisted exercise (Experimental): Robot-assisted exercise program will applied by patients with upper limb amputation using myoelectric prosthesis
  Interventions: Device: Robot
- Home exercise (Active Comparator): Home exercise program will applied by patients with upper limb amputation using myoelectric prosthesis
  Interventions: Other: Home exercise

INTERVENTIONS:
Device: Robot — Patients with upper limb amputation using myoelectric prosthesis will done robot-assisted exercise program
  Arms: robot-assisted exercise
Other: Home exercise — Patients with upper limb amputation using myoelectric prosthesis will done home exercise program
  Arms: Home exercise

SUMMARY:
The aim of this study was to investigate the effect of a robot-assisted biofeedback exercise program on grip strength, movement speed, coordination, functional status, depressive status, and quality of life in patients with a myoelectric prosthesis with upper limb amputation. In the literature review, There is no robot-assisted exercise program applied in patients using upper extremity myoelectric prosthesis.

The expected benefit from this study is to show that the functional status, depressive status, and quality of life of the patients who received robot-assisted biofeedback exercise were better than those who had a home exercise program only.

DETAILED DESCRIPTION:
The study was planned as a randomized prospective clinical study. The study was planned to include 16 patients. New amputation patients will be excluded from the study. The patients in the study group will have 5 sessions of exercise in the hospital for a week. The control group will receive a home exercise program.

Statistical analysis Student t-test will be used for the comparison of descriptive statistical methods (mean, standard deviation, median, frequency, and ratio) and normal distribution parameters between groups. Pearson chi-square test, Yates Continuity Correction, Fisher-Freeman-Halton Exact Test, Fisher Exact Test, and Marginal Homogeneity Test will be used to compare qualitative data. The results will be evaluated at 95 % confidence interval and p <0.01 and p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Upper elbow amputation
* Being using myoelectric prosthesis for amputated upper extremity
* Be literate
* To be able to complete and complete the tests at the level of mental and physical activity
* Being 18-65 years old

Exclusion Criteria:

* Patients with neurological sequelae
* Patients who could not cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Kinematic data | 1 day
  range of motion (ROM): unit is degree

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA AYDIN, MD, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Biffi E, Maghini C, Cairo B, Beretta E, Peri E, Altomonte D, Mazzoli D, Giacobbi M, Prati P, Merlo A, Strazzer S. Movement Velocity and Fluidity Improve after Armeo(R)Spring Rehabilitation in Children Affected by Acquired and Congenital Brain Diseases: An Observational Study. Biomed Res Int. 2018 Nov 18;2018:1537170. doi: 10.1155/2018/1537170. eCollection 2018. PMID 30581845
- [Derived] Aydin T, Kesiktas FN, Akbulut YD, Corum M, Ones K, Kizilkurt T, Bugdayci ND, Karacan I. The efficacy of robot-assisted training for patients with upper limb amputations who use myoelectric prostheses: a randomized controlled pilot study. Int J Rehabil Res. 2022 Mar 1;45(1):39-46. doi: 10.1097/MRR.0000000000000506. PMID 34775437